CLINICAL TRIAL: NCT04231799
Title: The Effect of Delayed First Bathing on Skin Barrier Function, Body Temperature and Comfort in Late Preterm Infants
Brief Title: Delaying First Bathing and Skin Barrier Function on Infant
Acronym: TEWL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Halil Ibrahim Tasdemir, Principal Investigator, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KAEK-30
Record Dates: First submitted 2020-01-09; First posted 2020-01-18 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Premature; Thermoregulation
Keywords: First Bathing; TEWL; Neonatal intensive care unit; Nursing care; Premature infant; Skin care; Comfort
MeSH Terms: conditions — Premature Birth | interventions — Baths

STUDY DESIGN:
Intervention Model Description: Randomized controlled multicenter double blind trial
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The person who will bathe the baby will not know the postnatal age of the baby. he will not know at what time of birth the baby's first bath is applied.
  The two assessors who will measure the results will not know the postnatal age of the baby and in which group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bathing within 24-48 (Experimental): Participants who will have their first bath in 24-48th hours after birth.
  Interventions: Procedure: Bathing
- Bathing within 48-72 (Experimental): Participants who will have their first bath in 48-72th hours after birth.
  Interventions: Procedure: Bathing

INTERVENTIONS:
Procedure: Bathing — Traditionally, it is the process of washing the newborn in the first hours of life to remove blood, meconium, varnish and other infectious substances.

SUMMARY:
It is still unknown when the first bath should be done in premature newborns. Investigators think that delaying the time of the first bath compared to the time in the clinic will show some positive changes in preterm newborns.

DETAILED DESCRIPTION:
Bath procedures and timing to reduce neonatal stress and protect the skin barrier should be preferred. This study aims to investigate the effect of delaying the first bath on skin barrier function, comfort and body temperature in late preterm infants. The study, between March 2020 and March 2021 in Turkey / Antalya will be held in three central provinces in the Neonatal Intensive Care Unit. Skincare is routinely performed between 08.00 and 09.00 in the form of a tub bath. This study sampled 80 stable, late preterm infants who were cared for in the NICU. This example was considered to be sufficient based on a sample size calculation in PS Power and Sample Size Calculations (Version 3.0). Allocations about the allocation were provided only by the lead researcher. Participants were given a sequential number placed in an opaque, closed envelope by the researcher who received the signed parental informed consent. When the participant is planned to take a bath, the researcher will be blind. The researcher who will apply the bathing process will not know the postnatal age of the baby when bathing. And the outcome evaluation of the participants was blinded. The participants were randomly divided into two groups. The bath will be applied to one group within the first 48 hours and the other group within 48-72 hours. The participants will then be placed in a preheated incubator that varies according to the weight and age of the participant. To compensate for such differences, the heads of all participants will be placed at a height of 30 degrees in the right lateral position after bathing. After the bath, participants were left without intervention or contact for about 10 minutes or until they settled before being evaluated. The participant Baths Work Record, a data collection tool, was designed specifically for this study. The instrument includes a series of scales for measuring outcome variables and demographic information (age, sex, mode of delivery, gestational age, birth weight, bodyweight at work, etc.). Outcome measurements include transepidermal water loss for skin barrier function, neonatal comfort behavior, and body temperature. Those responsible for data collection will be blinded in the allocation of the participants they evaluate. The ComfortNeo scale will be used to measure the comfort and pain intensity of newborns. The outcome criteria will be evaluated in three separate cases (10 minutes before bath, 1 minute and 10 minutes after bath). SPSS 20.0 and SAS (ver. 9.3) will be used and statistical significance will be set to p <0.05.

The data will be presented as means and standard deviations for continuous variables and as frequencies for categorical variables. For participant characteristics such as birth type and gender, the chi-square test will be used to determine whether there is a significant difference between the groups. Participant characteristics such as birth weight and body weight during the study will be evaluated for significant intergroup differences using a one-way ANOVA test. In order to compare different phases, the measurement parameters (comfort score, body temperature) in the baths will be averaged separately. To analyze both intra-group and intra-group differences, repeated variance analysis followed by Bonferroni's post hoc test.

ELIGIBILITY:
Inclusion Criteria:

* Born between 34 weeks + 0 days and 36 weeks + 6 days (late preterms),
* With a body weight of over 2000g,
* Spontaneous breathing,
* Preterms with stable physiological parameters

Exclusion Criteria:

* Receiving mechanical ventilation support,
* HIV, Hepatitis B mother baby,
* Preterms bathed before the intervention,
* Surgical procedure and incision in any region,
* Preterms with central catheters,
* Preterms with systemic infection,
* Preterms using sedative and / or muscle relaxants,
* Preterms with congenital, chromosomal abnormalities

Ages: 24 Hours to 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Skin Barrier Function | The Skin Barrier Function will be carried out by measuring trans epidermal water loss 10 minutes before first bath and 10 minutes after first bath.
  Transepidermal water loss of the participants will be measured using the VapoMeter SWL-2 ™ (Delfin Technologies Ltd). The skin barrier function of the participants will be evaluated in this way.

SECONDARY OUTCOMES:
Comfort | The comfort will be carried out by ComfortNeo scale 10 minutes before first bath, 1 minutes after first bath and 10 minutes after first bath.
  The ComfortNeo scale will be used to measure newborns' comfort. The ComfortNeo is a Likert-type scale consisting of six parameters: alertness, calmness/agitation, crying, body movement, facial tension, and (body) muscle tone. The lowest score that can be obtained using this scale is 6, and the highest score is 30. Scores in the range of 6 to 13 indicate that the newborn is comfortable, while scores 14-30 are indicative of pain or distress in the newborn, thus necessitating comforting.
Body temperature | The body temperature will be measured by digital thermometers 10 minutes before first bath, 1 minutes after first bath and 10 minutes after first bath.
  Axillary body temperature of infants

CONTACTS AND LOCATIONS:
Overall Officials: Emine EFE, Study Director — Akdeniz University Children's Health and the Nursing Department
Locations (1):
- Akdeniz Universty, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It is not yet decided. After the study was finalized, the decision was planned.

REFERENCES:
- [Background] Tasdemir HI, Efe E. The effect of tub bathing and sponge bathing on neonatal comfort and physiological parameters in late preterm infants: A randomized controlled trial. Int J Nurs Stud. 2019 Nov;99:103377. doi: 10.1016/j.ijnurstu.2019.06.008. Epub 2019 Jun 21. PMID 31442786
- [Derived] Tasdemir HI, Efe E. The effect of delaying first bathing on skin barrier function in late preterm infants: A study protocol for multi-centre, single-blind RCT. J Adv Nurs. 2021 Feb;77(2):1051-1061. doi: 10.1111/jan.14657. Epub 2020 Nov 18. PMID 33210328